CLINICAL TRIAL: NCT03522116
Title: Relationship Between CMR-derived Parameters of Ischemia / Reperfusion Injury and the Timing of CMR After Reperfused ST-segment Elevation Myocardial Infarction
Brief Title: Relationship Between CMR-derived Parameters of Ischemia / Reperfusion Injury and Timing of CMR in STEMI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Pier Giorgio Masci, MD, PhD, Centre Hospitalier Universitaire Vaudois
Other Study IDs: TimingReperfusionInjury
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This a prospective observational study including patients with ST-segment elevation myocardial infarction undergoing cardiovascular magnetic resonance for clinical reason during the index hospitalization. This local registry stemmed from multi-center european registry on cardiovascular magnetic resonance

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of STEMI
* Undergoing CMR during the index hospitalization

Exclusion Criteria:

* Refractory cardiogenic shock
* claustrophobia
* eGFR<30 ml/min/1.73m2

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted to Lausanne University Hospital with the diagnosis of STEMI
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Metrics of ischemia / repercussion injury | June 2017

IPD SHARING:
Plan to Share IPD: No